CLINICAL TRIAL: NCT01070901
Title: Evaluation of Predictors of Immune Status in Solid Organ Transplantation
Brief Title: Immune Status in Solid Organ Transplantation
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: PROG-9F09
Record Dates: First submitted 2010-02-17; First posted 2010-02-18 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Organ Transplants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Organ transplant recipients

SUMMARY:
Immunosuppressive therapy protocols in solid organ transplantation are rudimentary, differ by transplant center and no practical strategies are available to guide an individuals' response to immune suppression. In this study we will conduct research to assess immunologic status in solid organ transplant recipients, predicting immune reconstitution and outcomes after transplant to better guide the use of immunosuppressive medications.

ELIGIBILITY:
Inclusion Criteria:

* Impending kidney transplant
* Age >18
* Able to provide informed consent and comply with the study procedures

Exclusion Criteria:

* Age<18
* Concomitant illness, which by decision of investigator, may compromise the ability to perform this trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tranplant clinic population
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-05; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Immune Markers | 0, 3, 6, 9, 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States